CLINICAL TRIAL: NCT03266575
Title: Does Pulmonary Rehabilitation Improve Frailty and Sarcopenia in End Stage Liver Disease?
Brief Title: Pulmonary Rehabilitation in End-Stage Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000852
Record Dates: First submitted 2017-03-30; First posted 2017-08-30 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: End Stage Liver Disease
Keywords: Frailty; Sarcopenia; Pulmonary Rehabilitation
MeSH Terms: conditions — End Stage Liver Disease; Frailty; Sarcopenia

STUDY DESIGN:
Intervention Model Description: randomized to pulmonary rehab vs home based exercise rpogram
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary Rehabilitation (Active Comparator): Participants will participate in formal Pulmonary Rehabilitation Exercise program
  Interventions: Behavioral: Pulmonary Rehabilitation Exercise
- Home based program (Active Comparator): Participants will participate in a Home based Exercise program
  Interventions: Behavioral: Home Based Exercise

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation Exercise — Participants will undergo Pulmonary Rehabilitation exercise. Participants will perform endurance (treadmill or cycle ergometer), strength (weight resistance) and flexibility training twice a week for a period of an hour per session
  Arms: Pulmonary Rehabilitation
Behavioral: Home Based Exercise — Participants will undergo Home based exercise program consisting of strength and conditioning. Participants will perform REST for 10 minutes daily, increasing to 20 minutes daily, after the second week, in their home environment. The total duration of the intervention will be 12 weeks. Participants will be provided with pedometers, REST video and binder, with instructions on how to perform exercises, and resistance bands.
  Arms: Home based program

SUMMARY:
The purpose of this study is to assess the impact of exercise on sarcopenia and frailty. The exercise that will be performed in this study will include either pulmonary rehabilitation or a formal home based video strengthening program

DETAILED DESCRIPTION:
Participants will be randomized into two groups. The Pulmonary Rehabilitation group will undergo exercise under a supervised setting for a total duration of 12 weeks. Patients will perform endurance (treadmill or cycle ergometer), strength (weight resistance) and flexibility training twice a week for a period of an hour per session. Exercises will be supervised by physiotherapists or exercise physiologists. Compliance and performance will be monitored by the trainer. They will receive a pedometer for home use. The Home based program group will perform REST for 10 minutes daily, increasing to 20 minutes daily, after the second week, in their home environment. The total duration of the intervention will be 12 weeks. Patients will be provided with pedometers, REST video and binder, with instructions on how to perform exercises, and resistance bands.

ELIGIBILITY:
Inclusion Criteria:

* wait listed for liver transplantation with poor 6 MWT

Exclusion Criteria:

* age < 18 years
* recent hospitalization (within 14 days) due to decompensation, variceal bleeding in the previous 1 month
* large esophageal varices without primary prophylaxis
* active excessive alcohol intake (in the previous 3 months)
* current overt uncontrolled hepatic encephalopathy
* hepatopulmonary syndrome with uncontrolled hypoxia
* portopulmonary hypertension
* inability to perform exercise
* marked symptomatic comorbidities (cardiac, pulmonary, renal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk test | baseline, 3 months
  Participants will walk on a straight, flat surface for 6 minutes at a self-determined pace.

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly D Watt, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials